CLINICAL TRIAL: NCT02826382
Title: A Preliminary Evaluation of Uptake in Bone Metastases, Biodistribution and Excretion of the Novel Radiotracer [68Ga]P15-041 by PET/CT
Brief Title: Preliminary Evaluation of Uptake in Bone Metastases and Biodistribution of [68Ga]P15-041
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Five Eleven Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 511-0001-A
Record Dates: First submitted 2016-07-05; First posted 2016-07-11 (Estimated); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Prostate Cancer; Bone Metastases
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (2):
- Dynamic imaging group (Experimental): Dynamic imaging of suspected bone metastases with the investigation drug [68Ga]P15-041
  Interventions: Drug: [68Ga]P15-041
- Whole body dosimetry group (Experimental): Determination of human dosimetry of the investigation drug [68Ga]P15-041
  Interventions: Drug: [68Ga]P15-041

INTERVENTIONS:
Drug: [68Ga]P15-041 — Imaging by Positron Emission Tomography after injection of [68Ga]P15-041

SUMMARY:
A phase1 study to demonstrate [68Ga]P15-041 binding to bone metastases in prostate cancer and determination of human dosimetry.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed prostate cancer. known or suspected bone metastases referred for a clinical [99mTc]MDP scan

Exclusion Criteria:

* Estimated creatinine clearance (GFR) < 30 mL/min (calculated), history of hyperparathyroidism, • Inability to tolerate imaging procedures in the opinion of an investigator or treating physician, • Any current medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician investigator to be a condition that could compromise participant safety or successful participation in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Time course of uptake of [68Ga]P15-041 in bone metastases | 60 minutes post injection
  kinetics of [68Ga]P15-041 uptake in known or suspected bone metastases in prostate cancer
Time course of whole body distribution of [68Ga]P15-041 | 3 hours post injection
  whole body distribution of [68Ga]P15-041 used for human dosimetry determination

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States